CLINICAL TRIAL: NCT03354338
Title: Efficacy of Intensive Periodontal Therapy and Premedication With Oral Amoxicilline on Inflammatory Markers and Bacteremia in Patients With Chronic Periodontitis. A Randomized Controlled Trial.
Brief Title: Amoxicillin to Prevent Bacteria and Inflammatory Biomarkers After Intensive Periodontal Therapy
Acronym: AMX-Perio
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad El Bosque, Bogotá (Other)
Responsible Party: Principal Investigator, Luis Antonio Noriega Frontado, MSc (c) Dentistry Science, Universidad El Bosque, Bogotá
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UIBObosque
Record Dates: First submitted 2017-11-16; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Chronic Periodontitis; Bacteremia
Keywords: Periodontal disease; Bacteremia; Amoxicilline; Inflamatory markers
MeSH Terms: conditions — Chronic Periodontitis; Bacteremia; Periodontal Diseases | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: A triple-blind randomized controlled trial with 90 participants will be conducted. Participants will be assigned using block randomization in two groups and will received intensive periodontal therapy under local anaesthesia.
  Test group pre-medication with 2 gr of oral amoxicilline 1 hour before treatment.
  Control group with 2 gr of placebo 1 hour before treatment. Samples of blood will be taken at baseline (before treatment), immediately finished the treatment, 30 minutes later, after 24 hours, after seven days and on the day 30th to asses bacteremia and inflammatory markers
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, Investigator, Outcomes Assessor and Statistic. The treatment codes of the study were not accessible to the investigators and to the examiner until the data will be analyzed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Intensive Periodontal treatment and pre-medication with 2 gr of oral amoxicilline 1 hour before treatment
  Interventions: Drug: Amoxicillin
- PLACEBO (Placebo Comparator): Intensive Periodontal treatment with 2 gr of Placebo 1 hour before treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Intensive Periodontal treatment; Pre-medication with 2 gr of oral Amoxicillin 1 hour before treatment
  Other Names: Intensive Periodontal treatment
  Arms: Experimental Group
Other: Placebo — Intensive Periodontal treatment; Pre-medication with 2 gr of Placebo 1 hour before treatment
  Other Names: Intensive Periodontal treatment
  Arms: PLACEBO

SUMMARY:
There are not published studies evaluating the incidence, nature, magnitude and/or duration of bacteremia after periodontal treatment. The pre-surgical antibiotics have been studied particullary over Gram positive bacterial but not over gram negative bacterial and their secondary effects over the systemic pro-inflamation. Objective: to evaluate the efficacy of intensive periodontal therapy and pre-medication with oral amoxicilline on inflammatory bio-markers and the incidence, duration and magnitude of bacteremia in patients with chronic periodontitis.

DETAILED DESCRIPTION:
A randomized, triple-blind clinical trial with 90 participants will be conducted (age range18-65 years) with chronic periodontitis will be received and intensive periodontal therapy under local anaesthesia. Participants will be randomly assigned using block randomization in two groups. Test group premedication with 2 gr of oral amoxicilline 1 hour before periodontal treatment and control group with 2 gr of placebo 1 hour before treatment. High-sensitivity assays will be used to quantify serum concentrations of inflammatory marker (Interleukin (IL-1β), Interleukin 6, Tumour necrosis factor α, MCP 1, C Reactive Protein (CRP), plasma haemostatic (D-dimer), and von Willebrand factor antigen (r-WF:Ag).

Samples of blood will be taken at baseline (before treatment), inmediatly finished the treatment, 30 minutes and 1, seven and 30 days after treatment to asses bacteremia and inflammatory markers.

Bacterial isolation and identification: Bacterial colonies will be isolated on both selective and nonselective culture medium for aerobes and anaerobes bacteria. Sensitive Digital quantitative polymerase chain reaction will be used to quantify bacteria.

Concentrations of CPRus, inflammatory, haemostatic and endotellial cell activation markers will be quantified by high-sensitive enzyme liked inmunosorbent assays according to the manufacturer´s protocol. For each cytokine, comparisons between groups will be made by time. The levels of cytokines expressed in picograms will be transformed into international units for the statistical analysis.

In case it follows a normal distribution, an analysis of variance (ANOVA) for repeated measurements between groups with post hoc corrections made by Wilcoxon test will be used. In case it doesn´t follow a normal distribution, Non parametric test such as Friedman´s test will be used. Values of p<0.05 will be accepted as statiscally significant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic periodontitis (Ameriacam Academy of Periodontology 2015), having at least 2 teeth for quadrant with periodontal probing pockets depth ≥ 5 mm.

Exclusion Criteria:

* Pregnant and lactating women, Diabetes, hypertension, Obesity, Allergy to penicillin, consumption of systemic antimicrobial or anti-inflamatory drugs in the last 2 months, Autoimmune diseases, patients with medical conditions that required antibiotic premedication such as prosthetic heart valve replacement, skeletal joint replacement, previous history of infective endocarditis and history of rheumatic fever.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence bacteria "Change" | baseline (before treatment), immediately finished the treatment, 30 minutes later, after 24 hours, after seven days and on the day 30th
  absence or presence bacterial in blood
Change of Nature of the bacteria | baseline (before treatment), immediately finished the treatment, 30 minutes later, after 24 hours, after seven days and on the day 30th
  bacterial strain
Change of magnitude of bacteremia | baseline (before treatment), immediately finished the treatment, 30 minutes later, after 24 hours, after seven days and on the day 30th
  Colony forming units (CFU)
Duration of bacteremia | baseline (before treatment), immediately finished the treatment, 30 minutes later, after 24 hours, after seven days and on the day 30th
  Bacteremia´s minutes

SECONDARY OUTCOMES:
Change of levels of Interleukin | baseline, immediately finished the treatment, 30 minutes, 24 hours, 7 days and day 30th later
  Levels pg/ml
Change of C Reactive Protein (CRP) | baseline, immediately finished the treatment, 30 minutes, 24 hours, 7 days and day 30th later
  Levels mg/L
Change of levels of plasma haemostatic (D-dimer) | baseline, immediately finished the treatment, 30 minutes, 24 hours, 7 days and day 30th later
  Levels ng/ml
Change of von Willebrand factor antigen (r-WF:Ag) | baseline, immediately finished the treatment, 30 minutes, 24 hours, 7 days and day 30th later
  Levels ng/ml
Change of Pressure blood | baseline, immediately finished the treatment
  Millimeter of mercury (mmHg)
Change of Heart rate. | baseline, immediately finished the treatment
  Beats per Minute (BPM)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Antonio Noriega Frontado, MSc (c), Principal Investigator — El Bosque University
Locations (1):
- Luis Antonio Noriega Frontado, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Academy of Periodontology Task Force Report on the Update to the 1999 Classification of Periodontal Diseases and Conditions. J Periodontol. 2015 Jul;86(7):835-8. doi: 10.1902/jop.2015.157001. Epub 2015 May 27. No abstract available. PMID 26125117
- [Background] Arduino PG, Tirone F, Schiorlin E, Esposito M. Single preoperative dose of prophylactic amoxicillin versus a 2-day postoperative course in dental implant surgery: A two-centre randomised controlled trial. Eur J Oral Implantol. 2015 Summer;8(2):143-9. PMID 26021225
- [Background] Axelsson P, Nystrom B, Lindhe J. The long-term effect of a plaque control program on tooth mortality, caries and periodontal disease in adults. Results after 30 years of maintenance. J Clin Periodontol. 2004 Sep;31(9):749-57. doi: 10.1111/j.1600-051X.2004.00563.x. PMID 15312097
- [Background] Beck J, Garcia R, Heiss G, Vokonas PS, Offenbacher S. Periodontal disease and cardiovascular disease. J Periodontol. 1996 Oct;67(10 Suppl):1123-37. doi: 10.1902/jop.1996.67.10s.1123. PMID 8910831
- [Background] Castillo DM, Sanchez-Beltran MC, Castellanos JE, Sanz I, Mayorga-Fayad I, Sanz M, Lafaurie GI. Detection of specific periodontal microorganisms from bacteraemia samples after periodontal therapy using molecular-based diagnostics. J Clin Periodontol. 2011 May;38(5):418-27. doi: 10.1111/j.1600-051X.2011.01717.x. Epub 2011 Mar 11. PMID 21392048
- [Background] Cobb CM. Clinical significance of non-surgical periodontal therapy: an evidence-based perspective of scaling and root planing. J Clin Periodontol. 2002 May;29 Suppl 2:6-16. PMID 12010523
- [Background] D'Aiuto F, Parkar M, Nibali L, Suvan J, Lessem J, Tonetti MS. Periodontal infections cause changes in traditional and novel cardiovascular risk factors: results from a randomized controlled clinical trial. Am Heart J. 2006 May;151(5):977-84. doi: 10.1016/j.ahj.2005.06.018. PMID 16644317
- [Background] D'Aiuto F, Parkar M, Tonetti MS. Acute effects of periodontal therapy on bio-markers of vascular health. J Clin Periodontol. 2007 Feb;34(2):124-9. doi: 10.1111/j.1600-051X.2006.01037.x. Epub 2007 Jan 3. PMID 17214734
- [Background] Daly CG, Mitchell DH, Highfield JE, Grossberg DE, Stewart D. Bacteremia due to periodontal probing: a clinical and microbiological investigation. J Periodontol. 2001 Feb;72(2):210-4. doi: 10.1902/jop.2001.72.2.210. PMID 11288795
- [Background] Dayer MJ, Jones S, Prendergast B, Baddour LM, Lockhart PB, Thornhill MH. Incidence of infective endocarditis in England, 2000-13: a secular trend, interrupted time-series analysis. Lancet. 2015 Mar 28;385(9974):1219-28. doi: 10.1016/S0140-6736(14)62007-9. Epub 2014 Nov 18. PMID 25467569